CLINICAL TRIAL: NCT06812455
Title: Effect of RIVAroxaban in Reducing Radial Artery Occlusion Rate After Transradial Coronary Catheterization
Brief Title: Effect of RIVAroxaban in Radial Artery Occlusion Treatment After Cardiac Catheterization
Acronym: RIVA-RAO
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Matthaios Didagelos, Consultant Interventional Cardiologist, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 107/2025
Record Dates: First submitted 2025-02-02; First posted 2025-02-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Radial Artery Occlusion
Keywords: radial artery occlusion; complications; transradial; coronary catheterization; treatment
MeSH Terms: conditions — Arterial Occlusive Diseases | interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Patients with RAO that will receive Rivaroxaban
  Interventions: Drug: Rivaroxaban
- Control (No Intervention): Patients with RAO that will not receive any anticoagulation

INTERVENTIONS:
Drug: Rivaroxaban — Patients with RAO that will receive p.o. tabs Rivaroxaban 20 mg q.d.
  Arms: Intervention

SUMMARY:
The purpose of the RIVA-RAO study is to determine whether the use of Rivaroxaban is an effective treatment of radial artery occlusion (RAO) after cardiac catheterization (both angiography and PCI). This is a prospective, single-center, randomized controlled, open-label study that will randomize patients with RAO into two groups, one receiving Rivaroxaban and the other receiving no anticoagulation. RAO will be detected by radial artery ultrasound up to 24 hours after the procedure.

Study objectives:

Primary objective:

To evaluate the effect of treatment with Rivaroxaban, in patients (both symptomatic and asymptomatic) with RAO after a coronary catheterization procedure (both angiography and percutaneous coronary intervention-PCI), in improving patency rates of the radial artery at 4 weeks after the procedure, compared with no-anticoagulation treatment.

Secondary objectives:

To compare local access site and systemic complications (bleeding events, pseudoaneurysm, arteriovenous fistula) at 4 weeks after the procedure between the two groups.

DETAILED DESCRIPTION:
The use of the radial artery as an access site for coronary catheterization procedures, is constantly increasing because of lower rate of access site complications, shorter hospital stay, improved patient comfort and safer hemostasis. Radial artery occlusion remains a concern after transradial procedures, with a varied incidence, ranging from 5 to 38% as reported in the literature and probably reflecting different evaluation methods (pulse palpation versus ultrasound).

Although perceived as usually asymptomatic, RAO may be symptomatic in up to 58.8% of patients, presenting as pain in the forearm, numbness/ paresthesia, paresis or acute ischemia. Moreover RAO excludes the affected vessel from future catheterization procedures, hemodialysis shunts, invasive hemodynamic monitoring, coronary arterial bypass grafting.

Spontaneous recanalization of the vessel after RAO ranges from 5.4 to 47% at 1-month follow up. Today the only randomized studies reagrding RAO treatment have used either low-molecular-weight-heparin (LMWH) or apixaban.

This is a prospective, randomized study that will enroll, after informed written consent, all consecutive patients presenting with RAO, after a coronary catheterization procedure (both angiography and PCI) through the transradial access and having successfully received at least one radial artery sheath of any size at the end of the procedure.

RAO will be diagnosed by radial artery ultrasound (2D, Doppler, colour) performed in all patients after sheath removal and successful local hemostasis and before hospital discharge. Clinical evaluation of radial artery patency with pulse palpation, modified Allen's test and reverse Barbeau test will be also applied in all patients.

Patients diagnosed with RAO will be randomized 1:1 into two groups:

Treatment group, that will receive Rivaroxaban for 4 weeks. Control group, that will not receive any anticoagulation.

All patients with RAO will be re-evaluated by radial artery ultrasound at 1-, 2- 4- weeks to determine radial artery patency and record any bleeding complications according to the EASY (Early Discharge After Transradial Stenting of Coronary Arteries) Hematoma Classification and the BARC (Bleeding Academic Research Consortium) bleeding definition.

ELIGIBILITY:
Inclusion Criteria:

1. Patients (both male and female) undergoing a coronary catheterization procedure (both angiography and PCI) through the transradial access and having successfully received at least one radial artery sheath of any size at the end of the procedure
2. Radial artery occlusion confirmed by ultrasound (2D, Doppler, colour)

Exclusion Criteria:

1. Age < 18 years
2. Unable to provide informed written consent
3. Any contraindication to receive Rivaroxaban

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Radial artery patency | 4 weeks
  Radial artery patency at 4 weeks after the procedure, evaluated with radial artery ultrasound.

SECONDARY OUTCOMES:
Bleeding events | 4 weeks
  To compare bleeding events (based on the BARC bleeding definition) at 4 weeks after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Ziakas, Professor, Study Chair — AHEPA University Hospital, Thessaloniki, Greece
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amirpour A, Zavar R, Seifipour A, Sadeghi M, Shirvani E, Kermani-Alghoraishi M, Sanei H, Hashemi Jazi SM, Pourmoghaddas A, Khosravi Farsani A, Zarepour E, Safaei A, Hassannejad R. Apixaban, a Novel Oral Anticoagulant, Use to Resolute Arterial Patency in Radial Artery Occlusion Due to Cardiac Catheterization; A Pilot Randomized Clinical Trial. ARYA Atheroscler. 2023 Nov-Dec;19(6):18-26. doi: 10.48305/arya.2023.41915.2909. PMID 38883851
- [Background] Bernat I, Aminian A, Pancholy S, Mamas M, Gaudino M, Nolan J, Gilchrist IC, Saito S, Hahalis GN, Ziakas A, Louvard Y, Montalescot G, Sgueglia GA, van Leeuwen MAH, Babunashvili AM, Valgimigli M, Rao SV, Bertrand OF; RAO International Group. Best Practices for the Prevention of Radial Artery Occlusion After Transradial Diagnostic Angiography and Intervention: An International Consensus Paper. JACC Cardiovasc Interv. 2019 Nov 25;12(22):2235-2246. doi: 10.1016/j.jcin.2019.07.043. PMID 31753298
- [Background] Tsigkas G, Papanikolaou A, Apostolos A, Kramvis A, Timpilis F, Latta A, Papafaklis MI, Aminian A, Davlouros P. Preventing and Managing Radial Artery Occlusion following Transradial Procedures: Strategies and Considerations. J Cardiovasc Dev Dis. 2023 Jun 30;10(7):283. doi: 10.3390/jcdd10070283. PMID 37504539
- [Background] Didagelos M, Pagiantza A, Zegkos T, Papanastasiou C, Zarra K, Angelopoulos V, Kouparanis A, Peteinidou E, Sianos G, Karvounis H, Ziakas A. Low-molecular-weight heparin in radial artery occlusion treatment: the LOW-RAO randomized study. Future Cardiol. 2022 Feb;18(2):91-100. doi: 10.2217/fca-2021-0067. Epub 2021 Aug 16. PMID 34397270
- [Background] Didagelos M, Pagiantza A, Zegkos T, Zarra K, Angelopoulos V, Kouparanis A, Peteinidou E, Kassimis G, Karvounis H, Ziakas A. Low Molecular Weight Heparin in Improving RAO After Transradial Coronary Catheterization: The LOW-RAO Randomized Study. JACC Cardiovasc Interv. 2022 Aug 22;15(16):1686-1688. doi: 10.1016/j.jcin.2022.05.047. Epub 2022 Jul 27. No abstract available. PMID 35981848